CLINICAL TRIAL: NCT05330897
Title: A Multicentre Post Marketing Study in France Evaluating the Safety and Efficacy of the eCLIPs™ Family of Products for the Treatment of Bifurcation Intracranial Aneurysms at the Carotid and Basilar Terminus
Brief Title: French eCLIPs™ Efficacy and Safety Investigation
Acronym: EESIS-Fr
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evasc Medical Systems Corp. (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-15-015
Record Dates: First submitted 2022-03-10; First posted 2022-04-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Intracranial Aneurysm
Keywords: Bifurcation aneurysm; Basilar tip; Carotid terminus
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Implantation of an eCLIPs™ device
  Interventions: Procedure: Implantation of an eCLIPs™ device; Device: eCLIPs™ Electrolytic Bifurcation Systems

INTERVENTIONS:
Procedure: Implantation of an eCLIPs™ device — Implantation of an eCLIPs™ device and coiling of the bifurcation aneurysm
Device: eCLIPs™ Electrolytic Bifurcation Systems — Implantation of an eCLIPs™ device and coiling of the bifurcation aneurysm

SUMMARY:
The objective of this study is to demonstrate the safety and efficacy of the eCLIPs™ products for the treatment of bifurcation aneurysms.

DETAILED DESCRIPTION:
This study is a multicentre, open label, historically controlled, single-arm safety and efficacy study of the eCLIPs™ products in the management of bifurcated intracranial aneurysms at basilar tip and carotid terminus. Patients with basilar tip and carotid terminus aneurysms are not considered suitable for surgical treatment by the neurovascular community because of the poor outcome in these localizations. Patients included in the study will have saccular intracranial aneurysms that arise at or adjacent to a bifurcation, having a neck length of ≥ 4mm or have a dome:neck ratio <2. Efficacy will be measured as the proportion of aneurysms achieving complete occlusion (Raymond-Roy 1) at 12 months, while safety will be measured as the proportion of patients without a major stroke or non-accidental death within 30 days (procedural) and without a major ipsilateral stroke or neurological death between 31 days and 12 months. Additional endpoints will be evaluated and data collected to assess safety and collect information on the eCLIPs™ family of products.

ELIGIBILITY:
Inclusion Criteria:

1. Patient whose age is greater than 18 years old
2. Patient with an unruptured or previously ruptured (at least 1 month from date of rupture and with partial occlusion of the dome of the aneurysm by endovascular techniques or by open neurosurgery, and in stable neurological condition-WFNS I and II with a good recovery to at least to mRS 0-2) saccular, intracranial aneurysm or recurrent aneurysm, which arises at a bifurcation of Basilar Tip or Carotid Terminus with a minimal diameter of 5mm and a maximal diameter <25mm, has a neck length of >4mm or dome:neck ratio <2, branch artery diameters in the range of 2.0mm to 3.25mm
3. Patient aneurysm arises at a bifurcation artery with at least one of the two branch artery vessels having a diameter between 2.0mm and 3.25mm
4. Patient understands the nature of the procedure and has the capacity to provide informed consent (including fluency in French language)
5. Patient is willing to have on-site 30- day, 6-month, and 12 month follow-up evaluations as per standard clinical practice

Exclusion Criteria:

1. Patient with an aneurysm deemed to be an eligible candidate for surgical clipping by the investigator
2. Patient who presents with an intracranial mass or currently undergoing radiation therapy for carcinoma of the head or neck region
3. Major surgery within previous 30 days or planned in the next 120 days after enrolment
4. Patient with an International Normalized Ratio (INR) ≥ 1.5
5. Patient with serum creatinine level ≥104 µmol/L (or 2.5mg/dL) at time of enrolment
6. Patient with a platelet count ˂100x103 cells/mm3 or known platelet dysfunction at time of enrolment
7. Patient who has a known cardiac disorder, likely to be associated with cardio-embolic symptoms such as atrial fibrillation
8. Patient with any condition that, in the opinion of the treating physician, would place the participant at a high risk of embolic stroke or with any medical co-morbidity likely to affect the outcome (e.g. pulmonary disease, uncontrolled diabetes, blood disorders)
9. Patient with known allergies to nickel-titanium metal
10. Patient with known allergies to aspirin, heparin, ticlopidine, clopidogrel, prasugrel or other anti-platelet or P2Y12 agents or to general anesthesia
11. Subject has resistance to P2Y12 agents based on a validated platelet testing method (Verify Now, Multiplate or other)
12. Patient with a life threatening allergy to contrast (patients with itching or rash as a reaction to contrast can be included if properly prophylactically treated)
13. Patient with inappropriate anatomy as demonstrated by angiography due to severe intracranial vessel tortuosity or stenosis, or intracranial vasospasm not responsive to medical therapy
14. Patient who is currently participating in another clinical research study involving an investigational product
15. Patient who has had a previous intracranial procedure associated with the target aneurysm such that access and placement of an eCLIPs™ device would be compromised
16. Stenting, angioplasty, or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to the treatment date
17. More than one intracranial aneurysm that requires treatment within 12 months.
18. Asymptomatic extradural aneurysms requiring treatment
19. Severe neurological deficit that renders the subject incapable of living independently
20. Unstable neurological deficit (i.e. worsening or improvement of clinical condition in the last 30 days
21. Dementia or psychiatric problem that prevents the subject from completing required follow up
22. Subject had a subarachnoid haemorrhage within 1 month prior to enrolment date
23. Subject has a non-treated arterio-venous malformation in the territory of the target aneurysm
24. Subject has a need for long-term use of anticoagulants
25. Patient who is unable to complete the required follow-up
26. Inability to understand the study or history of non-compliance with medical advice
27. Evidence of active infection at the time of treatment
28. Patient who is pregnant or breastfeeding
29. Patient who has participated in a drug study within the last 30 days
30. Patient over the age of majority benefiting from legal protection (guardianship, curatorship, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Complete aneurysm occlusion with no recurrence or re-treatment | 12 months
  Percent of subjects with complete aneurysm occlusion with no recurrence or re-treatment
Major stroke or non-accidental death within 30 days, or major ipsilateral stroke or neurological death between 31 days and 12 months | 12 months
  Percent of subjects with a major stroke or non-accidental death within 30 days or with a major ipsilateral stroke or neurological death between 31 days and 12 months

SECONDARY OUTCOMES:
Technical success | Immediately after the procedure
  Proportion of successful eCLIPs™ device implants at the target aneurysm
Complete aneurysm occlusion | 24 months
  Percent of subjects with complete aneurysm occlusion at 6 and 24 months
Complete and nearly complete aneurysm occlusion | 24 months
  Percent of subjects with complete and nearly complete aneurysm occlusion at 6, 12 and 24 months
Major ipsilateral stroke or neurological death | 24 months
  Percent of subjects with a major ipsilateral stroke or neurological death
Success of adjuvant coiling into aneurysm after successful eCLIPs™ implant | Immediately after the procedure
  Proportion of subjects with procedural success for the ability to insert coils into the aneurysm beyond the successfully implanted eCLIPs™ device, and the eCLIPs™ device to satisfactorily retain coils
Modified Rankin Score | 24 months
  Percent of subjects experiencing deterioration of Rankin Score from baseline to 1 month, 6-month, 12-month, and 24-month follow-up
Serious Adverse Device Effects | 24 months
  Percent of subjects experiencing Serious Adverse Device Effects at 1, 6, 12 and 24 months
Unplanned aneurysm re-treatment | 24 months
  Percent of subjects having an unplanned aneurysm re-treatment within 12 or 24 months
Device migration | 24 months
  Proportion of device migration at 12 and 24 months
Artery stenosis | 24 months
  Measurement of artery stenosis by radiography at 6, 12 and 24 months
Artery patency | 24 months
  Qualitative assessment of artery patency at 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Blanc, MD, Principal Investigator — Hôpital Fondation Adolphe de Rothschild
Locations (28):
- France (28):
  - CHU d'Amiens, Amiens
  - Groupe Hospitalier Pellegrin, Bordeaux
  - CHRU de Brest - Hôpital Cavale Blanche, Brest
  - HCL - Hôpital Pierre Wertheimer, Bron
  - CHU de Caen Normandie, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CH de Colmar - Hôpital Louis Pasteur, Colmar
  - Clinique des Cèdres, Cornebarrieu
  - AP-HP - HU Henri-Mondor, Créteil
  - Hôpital François Mitterrand, Dijon
  - CHU Grenoble Alpes, Grenoble
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Limoges, Limoges
  - Hôpital de La Timone, Marseille
  - Hôpital privé Clairval, Marseille
  - CHU de Montpellier - Hôpital Guy de Chauliac, Montpellier
  - CHRU de Nancy - Hôpital Central, Nancy
  - CHU de Nice - Hôpital Pasteur, Nice
  - AP-HP - HU Pitié-Salpêtrière - Charles Foix, Paris
  - CH Sainte-Anne, Paris
  - Hôpital Fondation Adolphe de Rothschild, Paris
  - CHU de Poitiers, Poitiers
  - CHRU de Rennes -Hôpital Pontchaillou, Rennes
  - CHU de Rouen, Rouen
  - CHU de Nantes - Hôpital Laennec, Saint-Herblain
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHI Toulon, Toulon
  - CHRU de Tours - Bretonneau, Tours

REFERENCES:
- [Background] Fiorella D, Arthur AS, Chiacchierini R, Emery E, Molyneux A, Pierot L. How safe and effective are existing treatments for wide-necked bifurcation aneurysms? Literature-based objective performance criteria for safety and effectiveness. J Neurointerv Surg. 2017 Dec;9(12):1197-1201. doi: 10.1136/neurintsurg-2017-013223. Epub 2017 Aug 10. PMID 28798268